CLINICAL TRIAL: NCT01376479
Title: Phase I, Double Blind, Randomized, Placebo-controlled, Dose Escalation Study to Assess the Safety and Immunogenicity of a Prophylactic Vaccine Against Enterovirus Infection in Healthy Adults
Brief Title: Safety and Immunogenicity Study of an Inactivated Vaccine Against Hand, Foot and Mouth Disease Caused by Enterovirus 71
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inviragen Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: INV-EVR-101
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Hand, Foot and Mouth Disease
Keywords: HFMD; EV71; Enterovirus; INV21; Encephalitis
MeSH Terms: conditions — Hand, Foot and Mouth Disease; Enterovirus Infections; Encephalitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- INV21 Low Dose (Experimental)
  Interventions: Biological: INV21 Low Dose; Biological: Placebo
- INV21 High Dose (Experimental)
  Interventions: Biological: INV21 High Dose; Biological: Placebo

INTERVENTIONS:
Biological: INV21 Low Dose — Inactivated EV71 vaccine containing whole viral particles of EV71 formulated with aluminum hydroxide.
  Other Names: INV21
  Arms: INV21 Low Dose
Biological: INV21 High Dose — Inactivated EV71 vaccine consisting of whole viral particles of EV71 formulated with aluminum hydroxide.
  Other Names: INV21
  Arms: INV21 High Dose
Biological: Placebo — Phosphate Buffered Saline (PBS)

SUMMARY:
The purpose of this study is to evaluate the safety and immune response of an inactivated vaccine to prevent hand, foot and mouth disease (HFMD) caused by Enterovirus 71 (EV71).

DETAILED DESCRIPTION:
Hand, foot and mouth disease (HFMD) caused by Enterovirus 71 (EV71) can be severely debilitating for some children with a risk of paralysis and death. The most susceptible age group is the 1 to 5 year olds, and the disease is spread via the oral-fecal route. Currently, there is no antiviral therapy nor there is a vaccine available to prevent HFMD. In this study, an inactivated vaccine (INV21) based on the EV71 antigen will be evaluated in terms of safety and immune response that is generated after two doses of the vaccine are given to healthy adults. Safety assessments include the frequency and severity of systemic adverse events as well as local reactions. Immune response will be assessed by measurement of EV71 neutralizing antibody levels at specified time points throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 21 to 45 years, inclusive, at time of screening
* In good health as determined by medical history and physical examination.
* Normal clinical safety laboratory examinations.
* Body mass index (BMI) in the range 19-28 kg/m2.
* Documented negative serology for HIV, Hepatitis C antibody, and Hepatitis B surface antigen.
* Females of child bearing potential must have a negative urine pregnancy test result during screening and a negative urine pregnancy test immediately prior to vaccination.
* Willing and able to give written informed consent to participate.
* Willing and able to communicate with the Investigator and understand the requirements of the study.
* Low levels of EV71 neutralizing antibody.

Exclusion Criteria:

* Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent
* Clinically significant hematological (including bleeding disorders), renal, hepatic, pulmonary (including asthma), central nervous system (including epilepsy, seizures, convulsions, or chronic migraines), cardiovascular, or gastrointestinal disorders, according to Investigator's judgment.
* Ongoing rash or other dermatologic disease.
* Abnormal ECG as assessed by the Investigator.
* History of diabetes mellitus.
* Hypersensitivity to any vaccine.
* History of severe HFMD with CNS involvement.
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination.
* Planned receipt of any vaccine in the 4 weeks following each of the vaccinations in this study.
* History of thymic pathology, thymectomy, myasthenia or any immunodeficiency.
* History of recurring migraines or on prescription medication for treatment of recurring headaches or migraines.
* Positive urine test for drugs of abuse.
* Females who are pregnant or lactating

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Frequency of systemic adverse events and local reactions in healthy adults following two doses of INV21 given 28 days apart | 56 days
  Frequency and severity of systemic adverse events up to 56 days post first dose. Frequency and severity of local reactions up to 14 days post each dose.

SECONDARY OUTCOMES:
Immunogenicity of INV21 vaccine in healthy adults following two doses given 28 days apart | 8 months
  Geometric mean titers based on neutralizing antibody titers. Measurement of fold-increase over baseline of neutralizing titers against EV71. Durability of immune response at 2 months and 6 months after the last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Tambyah, MBBS, Principal Investigator — Department of Medicine, National University Hospital
Locations (1):
- Investigational Medicine Unit, National University Hospital, Singapore, Singapore